CLINICAL TRIAL: NCT02074995
Title: Multiple Ascending, Sequential, Placebo-controlled, Double-blind Study to Assess Safety, Tolerability and Efficacy of BVS857 in Severe Burn Subjects
Brief Title: Study of Tolerability and Efficacy of BVS857 in Severe Burn Subjects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was prematurely terminated due to recruitment issues
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CBVS857X2201
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Results first posted 2016-03-07 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Hypercatabolic Status Related to Severe Burn
Keywords: Burn, Severe burn, Lean body mass, Cachexia, Hypermetabolism, Catabolism, Wound healing
MeSH Terms: conditions — Burns; Cachexia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BVS857 Grp 1A open label (Experimental): 0.03 mg/kg of BVS857intravenously in open label manner
  Interventions: Biological: BVS857
- BVS857 Group 1B/1C, 2, 3, 4 Double Blind (Experimental)
  Interventions: Biological: BVS857
- Placebo Group 1B/1C, 2, 3, 4 (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Biological: BVS857 — Group 1A&1B receive first dose as IV then remaining doses as SC. Groups 2, 3 and 4 receive only SC doses.
  Arms: BVS857 Group 1B/1C, 2, 3, 4 Double Blind; BVS857 Grp 1A open label
Other: placebo — Group 1B receive first dose as IV then remaining doses as SC. Groups 2, 3 and 4 receive only SC doses.
  Arms: Placebo Group 1B/1C, 2, 3, 4

SUMMARY:
Study of tolerability and efficacy of BVS857 in severe burn subjects over 8 weeks and 15 weeks

DETAILED DESCRIPTION:
No formal analysis was performed as study was terminated due to low enrollment issues. (n=1 patient was enrolled)

ELIGIBILITY:
Inclusion Criteria:

* Burn injury comprising 2nd degree deep partial thickness and/or 3rd degree full thickness burns, ≥20% total body surface area with expected need for surgical intervention and not exceeding the sum of age plus burn size of 100 (Baux score)
* Dosing must occur within 8-12 days post-burn
* Subjects must weigh at least 45kgs (for group 1 with doses of 0.03mg/kg) and be under 100 kg to participate in the study

Exclusion Criteria:

* Spinal cord injury
* Hypoxic brain injury (Glasgow Coma Scale (GCS) <8) at screening
* True conductive electric burn with suspected neurologic injury
* Uncontrolled diabetes with HbA1c > 10% at screening, or known history of hypoglycemia,
* History of or active peripheral neuropathy or seizure disorder
* Systemic corticosteroids : > 10mg/d of prednisone or equivalent, other investigational treatments (excluding investigational dressings), medications for weight loss including megestrol acetate, androgens or oral beta agonists

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2014-02; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was planned to have 4 groups of patients. In Group 1: the bioavailability of BVS857 following subcutaneous administration was planned. Groups 2-4 (Group 4 optional) different BVS857 doses were planned for safety, PK and efficacy assessments. Study was terminated due to low enrollment as only 1 patient was enrolled
Groups:
- BVS857 Grp 1A Open Label: 0.03 mg/kg of BVS857 intravenously in open label manner followed by subsequent subcutaneous doses weekly at day 15,22 and 29.
Period: Overall Study
Arm/Group | BVS857 Grp 1A Open Label | Placebo Group 1B/1C, 2, 3, 4 | BVS857 Group 1B/1C, 2, 3, 4 Double Blind
Started | 1 | 0 | 0
Completed | 1 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | BVS857 Grp 1A Open Label
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events as a Measure of Safety and Tolerability
Description: Number of patients with adverse events as a measure of safety and tolerability
Time Frame: Over 1 year
Measure: Number; unit: Participants
Arm/Group | BVS857 Grp 1A Open Label
Number analyzed (Participants) | 1
Participants
  Adverse Events | 1
  Serious Adverse Events | 0
  Death | 0

2. Primary Outcome: Efficacy Measure by Change in Lean Body Mass (LBM)
Description: Total LBM is measured by dual energy X-ray absorptiometry (DXA) scan.
Time Frame: Groups 2,3&4: Baseline, Day 35, Day 85 and Day 106
Population: Terminated study underpowered due to low enrollment (n=1 patient). No analysis can be provided
Arm/Group | BVS857 Grp 1A Open Label
Number analyzed (Participants) | 0

3. Secondary Outcome: Serum Pharmacokinetics (PK) of BVS857: Cmax; The Observed Maximum Plasma (or Serum or Blood) Concentration Following Drug Administration
Time Frame: Groups 1: Day 1through to Day 56: Groups 2,3&4:Day 1 through to Day 105
Population: Terminated study underpowered due to low enrollment (n=1 patient). No analysis can be provided
Arm/Group | BVS857 Grp 1A Open Label
Number analyzed (Participants) | 0

4. Secondary Outcome: Serum Pharmacokinetics (PK) of BVS857: Tmax; The Time to Reach the Maximum Concentration After Drug Administration
Time Frame: Groups 1: Day 1through to Day 56: Groups 2,3&4:Day 1 through to Day 105
Population: Terminated study underpowered due to low enrollment (n=1 patient). No analysis can be provided
Arm/Group | BVS857 Grp 1A Open Label
Number analyzed (Participants) | 0

5. Secondary Outcome: Serum Pharmacokinetics (PK) of BVS857: AUClast; The Area Under the Plasma (or Serum or Blood) Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration
Time Frame: Groups 1: Day 1through to Day 56: Groups 2,3&4:Day 1 through to Day 105
Population: Terminated study underpowered due to low enrollment (n=1 patient). No analysis can be provided
Arm/Group | BVS857 Grp 1A Open Label
Number analyzed (Participants) | 0

6. Secondary Outcome: Serum Pharmacokinetics (PK) of BVS857: AUCinf; The Area Under the Plasma (or Serum or Blood) Concentration-time Curve From Time Zero to Infinity
Time Frame: Groups 1: Day 1through to Day 56: Groups 2,3&4:Day 1 through to Day 105
Population: Terminated study underpowered due to low enrollment (n=1 patient). No analysis can be provided
Arm/Group | BVS857 Grp 1A Open Label
Number analyzed (Participants) | 0

7. Secondary Outcome: Serum Pharmacokinetics (PK) of BVS857: T1/2; The Terminal Elimination Half-life
Time Frame: Groups 1: Day 1through to Day 56: Groups 2,3&4:ay D1 through to Day 105
Population: Terminated study underpowered due to low enrollment (n=1 patient). No analysis can be provided
Arm/Group | BVS857 Grp 1A Open Label
Number analyzed (Participants) | 0

8. Secondary Outcome: Serum Pharmacokinetics (PK) of BVS857: CL; The Systemic (or Total Body) Clearance From Plasma (or Serum or Blood) Following Intravenous Administration
Time Frame: Groups 1: Day 1through to Day 56: Groups 2,3&4:Day 1 through to Day 105
Population: Terminated study underpowered due to low enrollment (n=1 patient). No analysis can be provided
Arm/Group | BVS857 Grp 1A Open Label
Number analyzed (Participants) | 0

9. Secondary Outcome: Serum Pharmacokinetics (PK) of BVS857: Vz; The Volume of Distribution During the Terminal Elimination Phase Following Intravenous Administration
Time Frame: Groups 1: Day 1through to Day 56: Groups 2,3&4:Day 1 through to Day 105
Population: Terminated study underpowered due to low enrollment (n=1 patient). No analysis can be provided
Arm/Group | BVS857 Grp 1A Open Label
Number analyzed (Participants) | 0

10. Secondary Outcome: Serum Pharmacokinetics (PK) of BVS857: Vss; The Volume of Distribution at Steady State Following Intravenous Administration
Time Frame: Groups 1: Day 1through to Day 56: Groups 2,3&4:Day 1 through to Day 105
Population: Terminated study underpowered due to low enrollment (n=1 patient). No analysis can be provided
Arm/Group | BVS857 Grp 1A Open Label
Number analyzed (Participants) | 0

11. Secondary Outcome: Serum Pharmacokinetics (PK) of BVS857: Vz/F; The Apparent Volume of Distribution During the Terminal Elimination Phase Following Extravascular Administration
Time Frame: Groups 1: Day 1through to Day 56: Groups 2,3&4:Day 1 through to Day 105
Population: Terminated study underpowered due to low enrollment (n=1 patient). No analysis can be provided
Arm/Group | BVS857 Grp 1A Open Label
Number analyzed (Participants) | 0

12. Secondary Outcome: Serum Pharmacokinetics (PK) of BVS857: CL/F; The Apparent Systemic (or Total Body) Clearance From Plasma (or Serum or Blood) Following Extravascular Administration
Time Frame: Groups 1: Day 1through to Day 56: Groups 2,3&4:Day 1 through to Day 105
Population: Terminated study underpowered due to low enrollment (n=1 patient). No analysis can be provided
Arm/Group | BVS857 Grp 1A Open Label
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | BVS857 Grp 1A Open Label
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BVS857 Grp 1A Open Label (N=1)
bacteremia (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
Terminated study underpowered due to low enrollment (n=1 patient). No analysis can be provided

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety